CLINICAL TRIAL: NCT04819633
Title: Evaluation of Serum Sestrin Levels in Patients With Leiomyoma
Brief Title: Evaluating Serum Sestrin in Leiomyoma Patients
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nura Fitnat Topbas Selcuki, MD, Specialist in Obstetrics and Gynecology, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: Myomsestrin
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Uterine Leiomyoma
MeSH Terms: conditions — Myofibroma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: 30 patients within the reproductive ages (18-45 years) who were diagnosed with leiomyomas using transvaginal ultrasonography without any additional chronic, systemic or autoimmune disease, are not currently using any medical, hormonal, antiinflammatory treatments are included in this group.
  Interventions: Other: Determination of serum sestrin levels
- Control Group: 30 healthy subjects within the reproductive ages (18-45 years) who visited the outpatient gynecological clinic for routine examination who do not have any additional chronic, systemic or autoimmune disease, who are not currently using any medical, hormonal, antiinflammatory treatments are included in this group.
  Interventions: Other: Determination of serum sestrin levels

INTERVENTIONS:
Other: Determination of serum sestrin levels — Serum sestrin levels will be determined using venous blood samples obtained from the subjects.

SUMMARY:
Leiomyomas are the most common benign neoplasms of women's reproductive system affecting 20-30% of women within the reproductive ages. Sestrins are serum proteins which are highly expressed under circumstances of DNA damage, hypoxia and oxditive stress and play an important role in autophagia. The aim of this study is to evaluate the relationship of serum sestrin proteins with development of leiomyomas.

DETAILED DESCRIPTION:
Leiomyomas are the benign neoplasms of uterus and the role of genetics, estrogen levels and obesity has already been shown in their development. Higher levels of serum sestrin proteins have already been associated with DNA damage, hypoxia and oxidative stress and sestrin plays an important role in autophagia. In order to evaluate the role of serum sestrin in the development of leiomyomas 30 patients between 18-45 years of age who were diagnosed with uterine leiomyomas with transvaginal ultrasonography will be included in the study group. Their serum sestrin levels will be determined and compared with that of 30 healthy subjects recruited during the same study period at the same clinic.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age
* patients diagnosed with uterine leiomyomas will be included in the study group
* patients without any additional comorbidities
* patients without any autoimmune diseases

Exclusion Criteria:

* patients with systemic diseases
* patients with known chronic inflammatory diseases
* patients using hormonal and/or medical therapy
* pregnant women
* lactating women
* patients with malignant diseases

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since uterine leiomyomas are evaluated study will be conducted only with female patients
Study Population: 30 patients diagnosed with uterine leiomyomas within the above mentioned age group (reproductive ages) are included in the study group. 30 age matched healthy subjects are included in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Evaluating the role of autophagia in the development of leiomyomas by evaluating the serum sestrin levels. | 2 months
  Increased levels of serum sestrin proteins are associated with impaired autophagia. This association will be evaluated in the context of leiomyoma patients by measuring serum sestrin levels in blood samples obtained from these patients and comparing them with the sestrin levels measured in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Pinar Yalcin Bahat, MD, Study Director — University of Health Sciences Turkey, Istanbul Kanuni Sultan Suleyman Training and Research Hospital
Locations (1):
- Sisli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No